CLINICAL TRIAL: NCT00178984
Title: Biomagnetic Characterization of Gastric Dysrhythmias:Study 2
Acronym: SQUID
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Alan Bradshaw, Research Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 051175; 5R01DK058697 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Ischemia
Keywords: Blood supply; Mesentery
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- poor blood flow: Group with partial ischemia to the small intestine
- Good blood flow: Group with normal blood flow, given different conditions to effect electrical currents in normal smooth muscle

SUMMARY:
The purpose of this study is to use the Squid magnetometer (Superconducting QUantum Interference Device) to help diagnose electrical and mechanical abnormalities of the stomach and intestines.

DETAILED DESCRIPTION:
The Squid magnetometer is a non-invasive investigational device that measures the electrical activity in the smooth muscle of the intestines. Volunteers with normal bowel activity, those with gastric problems, and diabetics with gastric problems will be studied under the SQuid to determine normal and abnormal activity. Diabetics with an abnormal gastric emptying study will be asked to participate.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers, those with stomach problems, and Diabetics with abnormal gastric emptying study

Exclusion Criteria:

* Diabetics with a normal gastric emptying study
* Participants with claustrophobia

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care clinic
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2000-06; Primary Completion 2012-08-10 (Actual); Study Completion 2012-08-10 (Actual)

PRIMARY OUTCOMES:
to observe a difference in the magnetic activity between the normal and diseased smooth muscle of the stomach and intestines. | 2010

SECONDARY OUTCOMES:
to specifically study the electrical activity of diabetics with an abnormal gastric emptying. | 2010
Measurement of mesenteric ischemia | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Leonard A. Bradshaw, Ph.D., Principal Investigator — Vanderbilt University Department of Physics and Surgery
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States